CLINICAL TRIAL: NCT03362749
Title: Eastern Ablation Registry for Solid Tumor (EAST)
Acronym: EAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201703032RIND
Record Dates: First submitted 2017-05-22; First posted 2017-12-05 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumor Including Thyroid, Bone, Liver, Pancreas
MeSH Terms: interventions — Radiofrequency Ablation; Electroporation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RFA, MWA, cryo and IRE — local tumor ablation

SUMMARY:
Local tumor ablation is among the major anti-tumor modalities worldwide. Given the number of changes that have taken place in the field of tumor ablation in the past 10 years, it is our intention to ensure that this highly utilized standardization continues to remain relevant as it unites all investigators and clinicians practicing interventional oncology by providing a common language to describe therapies and outcomes, develop studies, and communicate with other medical specialties. In an attempt to attain greater Asian-wide adoption, the investigators will initiate the registry system for local tumor ablation in Taiwan, China, Korea, Singapore, Hong Kong and Thailand.

DETAILED DESCRIPTION:
Local tumor ablation is among the major anti-tumor modalities worldwide. Although surgical resection is potentially curative and beneficial to long-term patient survival, the majority of patients are deemed unresectable.

In 2003, the International Working Group on Image-Guided Tumor Ablation published a document titled "Image-Guided Tumor Ablation: Proposal for Standardization of Terms and Reporting Criteria". Ten years later, the field of tumor ablation continues to evolve. Tumor ablation modalities that were still being developed at the time of original preparation, such as microwave, irreversible electroporation (IRE), have been introduced and clinical niches are being defined. Preliminary clinical studies have matured into larger longer-term series with 5- and 10-year follow-up data on par with the surgical and medical oncology literature. Over the interim, our initial document has also given rise to several additional position statements within the field of interventional oncology and been the source for more focused societal statements on tumor ablation of liver, kidney, pancreas and musculoskeletal tumors.

Given the number of changes that have taken place in the field of tumor ablation in the past 10 years, it is our intention to ensure that this highly utilized standardization continues to remain relevant as it unites all investigators and clinicians practicing interventional oncology by providing a common language to describe therapies and outcomes, develop studies, and communicate with other medical specialties. In an attempt to attain greater Asian-wide adoption, the investigators will initiate the registry system for local tumor ablation in Taiwan, China, Korea, Singapore, Hong Kong and Thailand.

The main objective of the registry will be "improved precision and communication in this field that leads to more accurate comparison of technologies and results and ultimately to improved patient outcomes". This study aims to establish a local tumor ablation registry in Taiwan and collect real-life data regarding the safety, efficacy, changes in clinical presentation, and practice pattern of treatment in patients with clinically confirmed solid tumor including thyroid, bone, liver, pancreas and those which are scheduated to be treated by local tumor ablation including radiofrequency ablation, microwave ablation, cryoablation and irreversible electroporation The results collected from this registry and the analyses generated will be valuable reference for physicians in choosing treatment strategy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all inclusion criteria will be included:

  1. Males or non-pregnant females, at least 18 years of age (inclusive)
  2. Patients with clinically confirmed solid tumor including thyroid, bone, liver, pancreas and those which are scheduated to be treated by local tumor ablation including radiofrequency ablation, microwave ablation, cryoablation and irreversible electroporation
  3. Patients who have provided written informed consent
  4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
  5. American Society of Anaesthesiologists (ASA) score ≤ 3

Exclusion Criteria:

Patients who meet any exclusion criteria will be excluded:

1. The procedure of local ablation is not completed due to machine or patient problem
2. Received treatment with an investigational agent/ procedure within 30 days prior to local ablation
3. Known history of HIV infection
4. Women who are pregnant
5. Life expectancy is less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving local tumor ablation for solid tumor including thyroid, bone, liver, pancreas and those which are scheduated to be treated by local ablation including radiofrequency ablation, microwave ablation, cryoablation and irreversible electroporation will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
To observe the efficacy of local tumor ablation | through study completion, an average of 1 year
  Response rate (RR) to local tumor ablation

SECONDARY OUTCOMES:
The effect of local tumor ablation | up to 3 years
  time-to-progression
To observe the survival rate | up to 3 years
  overall survival (OS)
To observe the progression-free survival rate | up to 3 years
  to observe the progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, M.D. Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan